CLINICAL TRIAL: NCT01074918
Title: Potassium-Magnesium Citrate as a Blood Pressure Lowering Agent in Hypertensive Patients; Role of Natriuresis
Brief Title: Potassium-Magnesium Citrate as a Blood Pressure Lowering Agent in Hypertensive Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: none enrolled per PI
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Orson Moe, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 012007-080
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Pre-hypertension; Hypertension
Keywords: Pre-hypertension; Hypertension
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — potassium-magnesium citrate; Potassium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Potassium Magnesium Citrate (Experimental)
  Interventions: Drug: Potassium, Magnesium, Citrate
- Potassium Chloride (Active Comparator)
  Interventions: Drug: Potassium Chloride

INTERVENTIONS:
Drug: Potassium, Magnesium, Citrate — Potassium MAgnesium Citrate - 30 mEq potassium, 15 mEq Magnesium, 45 mEq Citrate in a powder mixture twice a day, mixed with a glass of water.
  Arms: Potassium Magnesium Citrate
Drug: Potassium Chloride — Potassium Chloride
  Arms: Potassium Chloride

SUMMARY:
The goal of this study is to compare the effects of Potassium Magnesium Citrate to Potassium Chloride on blood pressure among patients with pre-hypertension or mild hypertension. We will also test whether Potassium Magnesium Citrate increases excretion of large amounts of sodium in the urine.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 21 years
* BMI > 18.5 kg/m2 and < 40 kg/m2
* Prehypertension and mild hypertension: BP systolic 120-159 mmHg, diastolic 80-95 mmHg
* Must agree to limit lifestyle changes including: 1) embarking on a new exercise or weight reduction program 2) altering alcohol intake during the trial.

Exclusion Criteria:

* Taking blood pressure lowering medication
* Diabetes mellitus
* Renal disease
* Active cardiac disease
* Active liver disease
* Chronic diarrhea
* Chronic NSAID use
* Active or suspected drug use
* Uncontrolled psychiatric disease
* HIV infection
* Missed more than 20% of clinic visits in the last yr
* Prescription of diuretics for any reason
* A patient taking nutritional supplements including multivitamins that is unwilling to discontinue them,\
* Consumption of greater than 14 alcoholic beverages per week

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 8 weeks
  We have estimated to detect a 4 mmHg difference, with a standard deviation estimated at 8 mmHg.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dallas VA Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas